CLINICAL TRIAL: NCT01829945
Title: Study of the Relationships Between Apolipoprotein B-48 Kinetics and Expression of Genes That Regulate Intestinal Lipid Metabolism in Men With the Metabolic Syndrome.
Brief Title: Study of the Relationships Between Apolipoprotein B-48 Kinetics and Expression of Genes That Regulate Intestinal Lipid Metabolism in Men With the Metabolic Syndrome (SMB48)
Status: Completed | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Patrick Couture, MD, FRCP, PhD, Laval University
Other Study IDs: INAF-129-05-02
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Metabolic Syndrome X
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum Plasma Intestinal tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
Several lines of evidence indicate that a significant proportion of cardiovascular disease (CVD) events are attributable to the presence of a cluster of metabolic abnormalities and perturbations, defined as the metabolic syndrome. It has been estimated that approximately 25% of the North American adult population is living with the metabolic syndrome. Recent studies show that overaccumulation of atherogenic triglyceride-rich lipoproteins (TRL) seen in insulin-resistant patients is partly due to increased production rate of intestinally derived apolipoproteinB-48-containing lipoproteins. This is of interest because substantial evidence exists indicating that elevated levels of intestinal lipoproteins are associated with increased CVD risk. However, as indicated in the body of this grant proposal, the underlying mechanisms that lead to intestinal overproduction of lipoproteins in insulin-resistant states are poorly understood.

The general objective of the proposed research is to investigate the mechanisms by which the metabolic syndrome affects apolipoproteinB-48 secretion in human. The primary hypothesis is that insulin resistance will be associated with higher levels of intestinal lipoproteins because of an increased secretion of these particles.

ELIGIBILITY:
Inclusion Criteria:

Subjects with metabolic syndrome:

* Men aged between 18-60 years
* Waist circumference >102
* HDL-cholesterol < 1.1 mmol/L
* Triglycerides > 1.7 mmol/L
* Fasting blood glucose >6.1 mmol/L
* Normal blood pressure (<130/85)

Controls:

* Men aged between 18-60 years
* Waist circumference >102
* HDL-cholesterol > 1.1 mmol/L
* Triglycerides < 1.7 mmol/L
* Fasting blood glucose <6.1 mmol/L
* Normal blood pressure (<130/85)

Exclusion Criteria:

* Women
* Men < 18 or > 60 years
* Smokers (> 1 cigarette/day)
* Body weight variation > 10% during the last 6 months prior to the study baseline
* Subjects with a previous history of cardiovascular disease
* Subjects with Type 2 diabetes
* Subjects with a monogenic dyslipidemia
* Subjects on hypertension medications or medications known to affect lipoprotein metabolism or the integrity of gastrointestinal mucosa
* Subjects with endocrine or gastrointestinal disorders
* History of alcohol or drug abuse within the past 2 years
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: community sample
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change in TRL apolipoproteinB-48 production rate. | Week 1

SECONDARY OUTCOMES:
Changes in duodenal expression of genes that regulate intestinal lipid absorption. | Week 1
  Genes that regulate intestinal lipid absorption that will be measured are Niemann-Pick C1-like-1 (NPC1L1), Adenosine triphosphate(ATP)-binding cassette transporters (ABCG5/8), Fatty Acid Binding Protein (FABP), Sterol Regulatory Element Binding Protein (SREBP)
Change in duodenal expression of genes that regulate intestinal lipid synthesis. | Week 1
  Genes that regulate intestinal lipid synthesis that will be measured are Acyl-Coenzyme A (CoA): diacylglycerol acyltransferase (DGAT), Acyl-CoA:cholesterol O-transferase 2 (ACAT2) and 3-hydroxy-methylglutaryl-CoA reductase (HMG CoA reductase).
Change in synthesis of apolipoproteinB-48 containing lipoproteins (Microsomal triglyceride transfer protein (MTP), apolipoproteinB-48). | Week 1

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, FRCP, PhD, Principal Investigator — Laval University
Locations (1):
- Institute of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada